CLINICAL TRIAL: NCT00996892
Title: A Phase Ib, Open-Label, Dose-Escalation Study Evaluating the Safety, Tolerability and Pharmacokinetics of GDC-0973 in Combination With GDC-0941 When Administered in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Safety, Tolerability and Pharmacokinetics of Cobimetinib in Combination With Pictilisib in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A recommended Phase 2 dose and schedule was not identified and the study was terminated before initiation of Stage 2B.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEK4752g; GO01330 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-10-12; First posted 2009-10-16 (Estimated); Results first posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-11

CONDITIONS: Solid Tumors
Keywords: GDC0941; GDC0973; MEK; MEK Inhibitor; PI3K; PI3K Inhibitor; PI3 Kinase; PI3 Kinase Inhibitor
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — cobimetinib; 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine

ARMS (6):
- Dose Escalation Stage 1: Cobimetinib + Pictilisib (Experimental): Participants will receive cobimetinib capsules (at a starting dose of 20 milligrams [mg]) and pictilisib capsules (at a starting dose of 80 mg) from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Doses will be increased to identify maximum tolerated dose (MTD) or potential recommended Phase 2 dose (RP2D). Treatment will continue until disease progression, unacceptable toxicity, or any other discontinuation criterion meets.
  Interventions: Drug: Cobimetinib; Drug: Pictilisib
- Dose Escalation Stage 1A: Cobimetinib + Pictilisib (Experimental): Participants will receive cobimetinib capsules (at a starting dose of 100 mg) on Days 1, 4, 8, 11, 15, and 18 and pictilisib capsules (at a starting dose of 130 mg) from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Doses will be increased to identify MTD or potential RP2D.Treatment will continue until disease progression, unacceptable toxicity, or any other discontinuation criterion meets.
  Interventions: Drug: Cobimetinib; Drug: Pictilisib
- Dose Escalation Stage 1B: Cobimetinib + Pictilisib (Experimental): Participants will receive cobimetinib capsules (at a starting dose of 40 mg) and pictilisib capsules (at a starting dose of 130 mg) from Days 1 to 7 and then from Days 15 to 21 in continuous 28-day cycles. Participants will be off study drugs from Days 8 to 14 and from Days 22 to 28. Treatment will continue until disease progression, unacceptable toxicity, or any other discontinuation criterion meets.
  Interventions: Drug: Cobimetinib; Drug: Pictilisib
- Dose Expansion Stage 2: Cobimetinib + Pictilisib (Experimental): Participants will received cobimetinib capsules and pictilisib capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles, at doses identified as MTD/potential RP2D from Stage 1. Treatment will continue until disease progression, unacceptable toxicity, or any other discontinuation criterion meets. This indication specific cohort will include participants with Kirsten rat sarcoma viral oncogene homolog (KRAS) mutant non-small cell lung cancer (NSCLC); epidermal growth factor receptor (EGFR) T790M mutant and EGFR inhibitor-progressing NSCLC; pancreatic adenocarcinoma; and KRAS mutant colorectal cancer (CRC).
  Interventions: Drug: Cobimetinib; Drug: Pictilisib
- Dose Expansion Stage 2A: Cobimetinib + Pictilisib (Experimental): Participants received cobimetinib capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles, at doses identified as MTD/potential RP2D from Stage 1A. Treatment will continue until disease progression, unacceptable toxicity, or any other discontinuation criterion meets. This indication specific cohort will include participants with KRAS mutant NSCLC; EGFR T790M mutant and EGFR inhibitor-progressing NSCLC; pancreatic adenocarcinoma; KRAS mutant CRC, and KRAS mutant endometrioid carcinoma.
  Interventions: Drug: Cobimetinib; Drug: Pictilisib
- Dose Expansion Stage 2B: Cobimetinib + Pictilisib (Experimental): Participants will receive cobimetinib capsules and pictilisib capsules from Days 1 to 7 and then from Days 15 to 21 in continuous 28-day cycles, at doses identified as MTD/potential RP2D from Stage 1B. Participants will be off study drugs from Days 8 to 14 and from Days 22 to 28. Treatment will continue until disease progression, unacceptable toxicity, or any other discontinuation criterion meets. This indication specific cohort will include participants with KRAS mutant endometrioid carcinoma.
  Interventions: Drug: Cobimetinib; Drug: Pictilisib

INTERVENTIONS:
Drug: Cobimetinib — Repeated oral dosing.
  Other Names: GDC-0973; XL518
Drug: Pictilisib — Repeated oral dosing.
  Other Names: GDC-0941

SUMMARY:
This is an open-label, multicenter, Phase Ib dose-escalation study designed to assess the safety, tolerability and pharmacokinetics of oral dosing of cobimetinib and pictilisib administered in combination in patients with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, locally advanced or metastatic solid tumors for which standard therapy either does not exist or has proven ineffective or intolerable
* Evaluable disease or disease measurable per Response Evaluation Criteria in Solid Tumors (RECIST)
* Life expectancy greater than or equal to (>=) 12 weeks
* Adequate hematologic and end organ function
* Agreement to use an effective form of contraception for the duration of the study

Exclusion Criteria:

* History of prior significant toxicity from another mitogen-activated protein kinase (MEK) pathway inhibitor requiring discontinuation of treatment
* History of prior significant toxicity from another phosphoinositide 3-kinase (PI3K) pathway inhibitor requiring discontinuation of treatment
* Allergy or hypersensitivity to components of the cobimetinib or pictilisib formulations
* Palliative radiotherapy within 2 weeks prior to first dose of study drug treatment in Cycle 1
* Experimental therapy within 4 weeks prior to first dose of study drug treatment in Cycle 1
* Major surgical procedure or significant traumatic injury within 4 weeks prior to first dose of study drug treatment in Cycle 1, or anticipation of the need for major surgery during the course of study treatment
* Prior anti-cancer therapy within 28 days before the first dose of study drug treatment in Cycle 1
* History of diabetes requiring daily medication, or history of Grade >= 3 fasting hyperglycemia
* Current severe, uncontrolled systemic disease
* History of clinically significant cardiac or pulmonary dysfunction
* History of malabsorption or other condition that would interfere with enteral absorption
* Clinically significant history of liver disease (including cirrhosis), current alcohol abuse, or current known active infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus
* Any condition requiring anticoagulants, such as warfarin, heparin, or thrombolytics
* Active autoimmune disease
* Uncontrolled ascites requiring weekly large volume paracentesis for 3 consecutive weeks prior to enrollment
* Pregnancy, lactation, or breastfeeding
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms
* No other history of or ongoing malignancy that would potentially interfere with the interpretation of the pharmacodynamic or efficacy assays

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2009-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Chan, M.D., Ph.D., Study Director — Genentech, Inc.
Locations (5):
- United States (5):
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated before initiation of Stage 2B; hence Stage 2B cohorts were not applicable.
Groups:
- S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib: Stage 1 Cohort 1 (S1 C1): Participants received a single oral dose of pictilisib 80 milligrams (mg) capsules on Day 1 of Cycle 1 and a single oral dose of cobimetinib 20 mg capsules on Day 3 of Cycle 1, followed by continuous 21-day dosing with both cobimetinib and pictilisib at same doses from Days 8 to 28 and then 7 days off study drugs from Days 29 to 35 (Cycle 1 = 35 days). In subsequent cycles (28-day cycles), participants received 21-day dosing with both cobimetinib and pictilisib at same doses from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib: Stage 1 Cohort 2 (S1 C2): Participants received a single oral dose of pictilisib 100 mg capsules on Day 1 of Cycle 1 and a single oral dose of cobimetinib 20 mg capsules on Day 3 of Cycle 1, followed by continuous 21-day dosing with both cobimetinib and pictilisib at same doses from Days 8 to 28 and then 7 days off study drugs from Days 29 to 35 (Cycle 1 = 35 days). In subsequent cycles (28-day cycles), participants received 21-day dosing with both cobimetinib and pictilisib at same doses from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib: Stage 1 Cohort 3 (S1 C3): Participants received a single oral dose of pictilisib 80 mg capsules on Day 1 of Cycle 1 and a single oral dose of cobimetinib 40 mg capsules on Day 3 of Cycle 1, followed by continuous 21-day dosing with both cobimetinib and pictilisib at same doses from Days 8 to 28 and then 7 days off study drugs from Days 29 to 35 (Cycle 1 = 35 days). In subsequent cycles (28-day cycles), participants received 21-day dosing with both cobimetinib and pictilisib at same doses from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib: Stage 1 Cohort 4 (S1 C4): Participants received cobimetinib 40 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib: Stage 1 Cohort 5 (S1 C5): Participants received cobimetinib 40 mg capsules and pictilisib 130 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib: Stage 1 Cohort 6 (S1 C6): Participants received cobimetinib 60 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib: Stage 1 Cohort 6A (S1 C6A): Participants received cobimetinib 80 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib: Stage 1A Cohort A (S1A CA): Participants received cobimetinib 100 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 130 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib: Stage 1A Cohort B (S1A CB): Participants received cobimetinib 100 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib: Stage 1A Cohort C (S1A CC): Participants received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 130 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib: Stage 1A Cohort D (S1A CD): Participants received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib: Stage 1A Cohort E (S1A CE): Participants received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 245 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib: Stage 1A Cohort F (S1A CF): Participants received cobimetinib 150 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib: Stage 1A Cohort G (S1A CG): Participants received cobimetinib 150 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 245 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib: Stage 1B Cohort AX (S1B CAX): Participants received cobimetinib 40 mg capsules and pictilisib 130 mg capsules from Days 1 to 7 and then from Days 15 to 21 in continuous 28-day cycles. Participants were off study drugs from Days 8 to 14 and from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib: Stage 1B Cohort BX (S1B CBX): Participants received cobimetinib 40 mg capsules and pictilisib 180 mg capsules from Days 1 to 7 and then from Days 15 to 21 in continuous 28-day cycles. Participants were off study drugs from Days 8 to 14 and from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib: Stage 1B Cohort CX (S1B CCX): Participants received cobimetinib 60 mg capsules and pictilisib 130 mg capsules from Days 1 to 7 and then from Days 15 to 21 in continuous 28-day cycles. Participants were off study drugs from Days 8 to 14 and from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib: Stage 1B Cohort DX (S1B CDX): Participants received cobimetinib 60 mg capsules and pictilisib 180 mg capsules from Days 1 to 7 and then from Days 15 to 21 in continuous 28-day cycles. Participants were off study drugs from Days 8 to 14 and from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib: Stage 2 (S2) expansion cohort: Participants received cobimetinib 40 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. This indication specific cohort included participants with Kirsten rat sarcoma viral oncogene homolog (KRAS) mutant non-small cell lung cancer (NSCLC); epidermal growth factor receptor (EGFR) T790M mutant and EGFR inhibitor-progressing NSCLC; pancreatic adenocarcinoma; and KRAS mutant colorectal cancer (CRC).
- S2A Expansion: 125 mg Cobimetinib + 180 mg Pictilisib: Stage 2A (S2A) expansion cohort: Participants received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. This indication specific cohort included participants with KRAS mutant NSCLC; EGFR T790M mutant and EGFR inhibitor-progressing NSCLC; pancreatic adenocarcinoma; KRAS mutant CRC, and KRAS mutant endometrioid carcinoma.
Period: Dose-Escalation Stage 1
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib | S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib | S2A Expansion: 125 mg Cobimetinib + 180 mg Pictilisib
Started | 4 | 3 | 3 | 9 | 11 | 10 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 3 | 9 | 11 | 10 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 2 | 2 | 3 | 4 | 10 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose-Escalation Stage 1A
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib | S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib | S2A Expansion: 125 mg Cobimetinib + 180 mg Pictilisib
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 4 | 7 | 9 | 8 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 4 | 7 | 9 | 8 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 5 | 7 | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose-Escalation Stage 1B
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib | S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib | S2A Expansion: 125 mg Cobimetinib + 180 mg Pictilisib
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 3 | 5 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 3 | 5 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 3 | 3 | 0 | 0
Period: Expansion Stage 2
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib | S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib | S2A Expansion: 125 mg Cobimetinib + 180 mg Pictilisib
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 0
Period: Expansion Stage 2A
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib | S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib | S2A Expansion: 125 mg Cobimetinib + 180 mg Pictilisib
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 45
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 45
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- All Participants: All participants who received cobimetinib and pictilisib in any dose combination until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
Arm/Group | All Participants
Number analyzed (Participants) | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12.0)
Gender [Count of Participants; unit: Participants]
  Female | 109
  Male | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) During Dose Escalation Stages 1, 1A and 1B
Description: DLT was defined as 1 of the following toxicities considered treatment related by Investigator: Grade ≥3 non-hematologic, non-hepatic organ toxicity, excluding the following: Grade 3 nausea, vomiting, or diarrhea that resolved to Grade ≤1 within 7 days, Grade 3 rash or Grade ≥3 fatigue that resolved to Grade ≤2 within 7 days, Grade ≥3 hyperglycemia or lipid profile results that occurred during non-fasting conditions, Grade 3 or 4 elevation of serum creatine phosphokinase levels or Grade 3 non clinically significant (as assessed by Investigator) laboratory abnormality that was asymptomatic; Grade ≥3 febrile neutropenia; Grade ≥4 neutropenia (absolute neutrophil count <500/microliter) lasting >5 days; Grade ≥4 thrombocytopenia lasting >48 hours; Grade ≥4 anemia; Grade ≥3 total bilirubin, hepatic transaminase, alkaline phosphatase, lasting >72 hours; Grade ≥2 diffusion capacity of the lung for carbon monoxide concomitant with an absolute decrease of ≥20 percentage points from baseline.
Time Frame: Cohorts 1-3: Day 1 to Day 35, All other cohorts: Day 1 to Day 28
Population: Safety-evaluable population included all participants who received at least one dose of study drug. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: participants
Groups:
- S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib: Participants received a single oral dose of pictilisib 80 mg capsules on Day 1 of Cycle 1 and a single oral dose of cobimetinib 20 mg capsules on Day 3 of Cycle 1, followed by continuous 21-day dosing with both cobimetinib and pictilisib at same doses from Days 8 to 28 and then 7 days off study drugs from Days 29 to 35 (Cycle 1 = 35 days). In subsequent cycles (28-day cycles), participants received 21-day dosing with both cobimetinib and pictilisib at same doses from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib: Participants received a single oral dose of pictilisib 100 mg capsules on Day 1 of Cycle 1 and a single oral dose of cobimetinib 20 mg capsules on Day 3 of Cycle 1, followed by continuous 21-day dosing with both cobimetinib and pictilisib at same doses from Days 8 to 28 and then 7 days off study drugs from Days 29 to 35 (Cycle 1 = 35 days). In subsequent cycles (28-day cycles), participants received 21-day dosing with both cobimetinib and pictilisib at same doses from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib: Participants received a single oral dose of pictilisib 80 mg capsules on Day 1 of Cycle 1 and a single oral dose of cobimetinib 40 mg capsules on Day 3 of Cycle 1, followed by continuous 21-day dosing with both cobimetinib and pictilisib at same doses from Days 8 to 28 and then 7 days off study drugs from Days 29 to 35 (Cycle 1 = 35 days). In subsequent cycles (28-day cycles), participants received 21-day dosing with both cobimetinib and pictilisib at same doses from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib: Participants received cobimetinib 40 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib: Participants received cobimetinib 40 mg capsules and pictilisib 130 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib: Participants received cobimetinib 60 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib: Participants received cobimetinib 80 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib: Participants received cobimetinib 100 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 130 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib: Participants received cobimetinib 100 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib: Participants received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 130 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib: Participants received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib: Participants received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 245 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib: Participants received cobimetinib 150 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib: Participants received cobimetinib 150 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 245 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib: Participants received cobimetinib 40 mg capsules and pictilisib 130 mg capsules from Days 1 to 7 and then from Days 15 to 21 in continuous 28-day cycles. Participants were off study drugs from Days 8 to 14 and from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib: Participants received cobimetinib 40 mg capsules and pictilisib 180 mg capsules from Days 1 to 7 and then from Days 15 to 21 in continuous 28-day cycles. Participants were off study drugs from Days 8 to 14 and from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib: Participants received cobimetinib 60 mg capsules and pictilisib 130 mg capsules from Days 1 to 7 and then from Days 15 to 21 in continuous 28-day cycles. Participants were off study drugs from Days 8 to 14 and from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib: Participants received cobimetinib 60 mg capsules and pictilisib 180 mg capsules from Days 1 to 7 and then from Days 15 to 21 in continuous 28-day cycles. Participants were off study drugs from Days 8 to 14 and from Days 22 to 28. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3 | 9 | 11 | 10 | 4 | 3 | 3 | 4 | 7 | 9 | 8 | 5 | 4 | 3 | 3 | 5
participants | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1

2. Primary Outcome: Maximum Tolerated Combination Doses of Cobimetinib and Pictilisib During Dose-Escalation Stages 1, 1A and 1B
Description: MTD was determined (by Investigator) based on the DLTs, as well as adverse events (AEs) in dose-escalation Stages 1, 1A, and 1B that did not meet protocol-defined DLT criteria but indicated intolerability of a given dose combination. Separate combination MTDs were determined for each dose-escalation stage. DLT was defined as 1 of the following toxicities considered treatment related by Investigator: Grade ≥3 non-hematologic, non-hepatic organ toxicity; Grade ≥3 febrile neutropenia; Grade ≥4 neutropenia (absolute neutrophil count <500/microliter) lasting >5 days; Grade ≥4 thrombocytopenia lasting >48 hours; Grade ≥4 anemia; Grade ≥3 total bilirubin, hepatic transaminase, alkaline phosphatase, lasting >72 hours; Grade ≥2 diffusion capacity of the lung for carbon monoxide concomitant with an absolute decrease of ≥20 percentage points from baseline.
Time Frame: Cohorts 1-3: Day 1 to Day 35, All other cohorts: Day 1 to Day 28
Population: Safety-evaluable population. Here, number of participants analyzed = participants who were evaluable for this outcome and n = participants evaluable for specified categories.
Measure: Number; unit: mg
Groups:
- All Participants - Stages 1, 1A, 1B: All participants who received cobimetinib and pictilisib in any dose combination during Stages 1, 1A, and 1B, until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
Arm/Group | All Participants - Stages 1, 1A, 1B
Number analyzed (Participants) | 98
mg
  Stage 1: Cobimetinib (n = 44) | 40
  Stage 1: Pictilisib (n = 44) | 100
  Stage 1A: Cobimetinib (n = 34) | 125
  Stage 1A: Pictilisib (n = 34) | 180
  Stage 1B: Cobimetinib (n = 20) | NA — MTD for Stage 1B was not determined as the study was terminated prior to initiation of Stage 2B.
  Stage 1B: Pictilisib (n = 20) | NA — MTD for Stage 1B was not determined as the study was terminated prior to initiation of Stage 2B.

3. Primary Outcome: Time of Maximum Concentration (Tmax) of Cobimetinib on Day 3 - Stage 1, Cohorts 1-3
Time Frame: 0-4 hours pre-cobimetinib (Pr-C) dose, 0.5, 2, 4, 6 hours post-cobimetinib (Po-C) dose on Day 3, Day 4
Population: Pharmacokinetic (PK) population included all participants who had at least one cobimetinib and pictilisib plasma concentration available. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3
hours | 4.00 [2.0 to 4.0] | 4.00 [4.0 to 4.0] | 2.00 [2.0 to 2.0]

4. Primary Outcome: Maximum Plasma Concentration (Cmax) of Cobimetinib on Day 3 - Stage 1, Cohorts 1-3
Time Frame: 0-4 hours Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Day 3, Day 4
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3
nanograms per milliliter (ng/mL) | 27.6 (95) | 16.6 (78) | 97.0 (63)

5. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to 24 Hours Post-Dose (AUC0-24) of Cobimetinib on Day 3 - Stage 1, Cohorts 1-3
Time Frame: 0-4 hours Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Day 3, Day 4
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nonograms*hour per milliliter (ng*h/mL)
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3
nonograms*hour per milliliter (ng*h/mL) | 392 (88) | 279 (75) | 1190 (53)

6. Primary Outcome: Tmax of Pictilisib on Day 1 - Stage 1, Cohorts 1-3
Time Frame: 0-4 hours pre-pictilisib (Pr-P) dose, 0.5, 2, 4, 6 hours post-pictilisib (Po-P) dose on Day 1, Day 2, 0-4 hours Pr-C dose on Day 3
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3
hours | 3.00 [2.0 to 24.0] | 4.00 [2.0 to 4.0] | 2.00 [2.0 to 2.0]

7. Primary Outcome: Cmax of Pictilisib on Day 1 - Stage 1, Cohorts 1-3
Time Frame: 0-4 hours Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Day 1, Day 2, 0-4 hours Pr-C dose on Day 3
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3
ng/mL | 162 (37) | 185 (27) | 280 (41)

8. Primary Outcome: AUC0-24 of Pictilisib on Day 1 - Stage 1, Cohorts 1-3
Time Frame: 0-4 hours Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Day 1, Day 2, 0-4 hours Pr-C dose on Day 3
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3
ng*h/mL | 1680 (16) | 1950 (50) | 2680 (83)

9. Secondary Outcome: Tmax of Cobimetinib on Cycle 1 Day 1 (Cycle 1 Day 8 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: Cohorts 1-3: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 8, Cycle 1 Days 9, 15, 21; Cohorts 4-6A: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Day 2, 8, 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 11 | 10 | 4
hours | 4.00 [2.0 to 4.0] | 4.00 [2.0 to 24] | 2.00 [2.0 to 2.0] | 2.00 [2.0 to 4.0] | 2.00 [2.0 to 2.0] | 4.00 [2.0 to 4.0] | 3.00 [2.0 to 4.0]

10. Secondary Outcome: Cmax of Cobimetinib on Cycle 1 Day 1 (Cycle 1 Day 8 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: as for outcome 9
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 11 | 10 | 4
ng/mL | 20.2 (100) | 17.7 (62) | 87.4 (73) | 101 (63) | 61.0 (45) | 131 (66) | 138 (61)

11. Secondary Outcome: AUC0-24 of Cobimetinib on Cycle 1 Day 1 (Cycle 1 Day 8 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: Cohorts 1-3: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 8, Cycle 1 Days 9; Cohorts 4-6A: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Day 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 11 | 10 | 4
ng*h/mL | 299 (62) | 311 (53) | 1320 (56.6) | 1300 (61) | 957 (42) | 2050 (71) | 1790 (56)

12. Secondary Outcome: Tmax of Cobimetinib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: Cohorts 1-3: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 28, Cycle 1 Day 29, Cycle 2 Days 1, 15, 21; Cohorts 4-6A: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 21, Cycle 1 Day 22, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 9 | 3 | 1
hours | 6.00 [2.0 to 6.0] | 4.00 [4.0 to 6.0] | 2.00 [2.0 to 24] | 2.00 [2.0 to 4.0] | 4.00 [2.0 to 24] | 3.0 [2.0 to 24] | 4 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable.

13. Secondary Outcome: Cmax of Cobimetinib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: as for outcome 12
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 9 | 3 | 1
ng/mL | 37.1 (5.6) | 52.2 (57) | 228 (120) | 167 (56) | 138 (63) | 245 (79) | 87.4 (NA) — Measure dispersion not applicable as only one participant was evaluable.

14. Secondary Outcome: AUC0-24 of Cobimetinib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: Cohorts 1-3: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 28, Cycle 1 Day 29; Cohorts 4-6A: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 9 | 3 | 1
ng*h/mL | 749 (1.4) | 900 (70) | 4130 (94) | 2410 (66) | 2460 (57) | 4050 (110) | 1120 (NA) — Measure dispersion not applicable as only one participant was evaluable.

15. Secondary Outcome: Terminal Half-life (t1/2) of Cobimetinib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Description: Half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 12
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 9 | 3 | 1
hours | 49.3 [41 to 60] | 37.9 [32 to 43] | 31.7 [22 to 48] | 34.1 [32 to 37] | 43.2 [34 to 56] | 45.7 [41 to 56] | 40.5 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable.

16. Secondary Outcome: Apparent Clearance (CL/F) of Cobimetinib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: as for outcome 12
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/hr)
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 9 | 3 | 1
Liters per hour (L/hr) | 26.7 (1.4) | 22.2 (70) | 9.67 (94) | 16.6 (66) | 16.2 (61) | 14.8 (110) | 53.6 (NA) — Measure dispersion not applicable as only one participant was evaluable.

17. Secondary Outcome: Accumulation Ratio of Cobimetinib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Description: Accumulation ratio was calculated as: AUC0-24 at Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) divided by AUC0-24 at Cycle 1 Day 1 (Cycle 1 Day 8 for Cohorts 1-3).
Time Frame: Cohorts 1-3: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Days 8 and 28, Cycle 1 Days 9, 29; Cohorts 4-6A: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Days 1 and 21, Cycle 1 Days 2, 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 9 | 3 | 1
ratio | 2.51 (63) | 2.89 (43) | 3.14 (73) | 2.03 (36) | 2.90 (73) | 2.83 (54) | 1.77 (NA) — Measure dispersion not applicable as only one participant was evaluable.

18. Secondary Outcome: Tmax of Pictilisib on Cycle 1 Day 1 (Cycle 1 Day 8 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: Cohorts 1-3: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 8, Cycle 1 Day 9, 15, 21; Cohorts 4-6A: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Day 2, 8, 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 11 | 10 | 4
hours | 2.00 [2.0 to 4.0] | 2.00 [2.0 to 4.0] | 2.00 [2.0 to 2.0] | 2.00 [0.5 to 4.0] | 2.00 [2.0 to 4.0] | 2.00 [0.5 to 4.0] | 2.00 [2.0 to 4.0]

19. Secondary Outcome: Cmax of Pictilisib on Cycle 1 Day 1 (Cycle 1 Day 8 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: as for outcome 18
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 11 | 10 | 4
ng/mL | 196 (20) | 193 (16) | 329 (26) | 390 (60) | 302 (34) | 272 (54) | 355 (83)

20. Secondary Outcome: AUC0-24 of Pictilisib on Cycle 1 Day 1 (Cycle 1 Day 8 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: Cohorts 1-3: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 8, Cycle 1 Day 9; Cohorts 4-6A: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Day 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 11 | 10 | 4
ng*h/mL | 1660 (28) | 2150 (43) | 2600 (28) | 3360 (43) | 2770 (43) | 2870 (48) | 3240 (68)

21. Secondary Outcome: Tmax of Pictilisib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: Cohorts 1-3: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 28, Cycle 1 Day 29, Cycle 2 Days 1, 15, 21; Cohorts 4-6A: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 21, Cycle 1 Day 22, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 8 | 3 | 1
hours | 2.00 [2.0 to 6.0] | 2.00 [2.0 to 2.0] | 2.00 [2.0 to 4.0] | 2.00 [0.5 to 4.0] | 2.00 [2.0 to 6.0] | 2.00 [2.0 to 24] | 2.00 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable.

22. Secondary Outcome: Cmax of Pictilisib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: as for outcome 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 8 | 3 | 1
ng/mL | 198 (38) | 278 (100) | 459 (20) | 409 (49) | 374 (69) | 396 (48) | 441 (NA) — Measure dispersion not applicable as only one participant was evaluable.

23. Secondary Outcome: AUC0-24 of Pictilisib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Time Frame: Cohorts 1-3: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 28, Cycle 1 Day 29; Cohorts 4-6A: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 8 | 3 | 1
ng*h/mL | 2500 (21) | 2930 (150) | 5500 (34) | 3890 (63) | 4320 (58) | 4510 (40) | 4070 (NA) — Measure dispersion not applicable as only one participant was evaluable.

24. Secondary Outcome: t1/2 of Pictilisib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Description: Half-life is the time measured for the plasma concentration to decrease by one half. As planned, summary statistics were not derived if fewer than 3 participants had available data; however, if the number of participants analyzed = 1, then the observed data of the single participant was reported as geometric mean.
Time Frame: as for outcome 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 1 | 0 | 0 | 2 | 8 | 3 | 0
hours | 25.8 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable. |  |  | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data. | 24.7 [22 to 30] | 27.7 [22 to 41] |

25. Secondary Outcome: CL/F of Pictilisib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Description: as for outcome 16
Time Frame: as for outcome 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 8 | 3 | 1
L/hr | 32.0 (21) | 34.1 (150) | 14.5 (34) | 25.7 (63) | 30.1 (58) | 22.2 (40) | 24.6 (NA) — Measure dispersion not applicable as only one participant was evaluable.

26. Secondary Outcome: Accumulation Ratio of Pictilisib on Cycle 1 Day 21 (Cycle 1 Day 28 for Cohorts 1-3) - Stage 1 All Cohorts
Description: as for outcome 17
Time Frame: Cohorts 1-3: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Days 8 and 28, Cycle 1 Days 9, 29; Cohorts 4-6A: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Days 1 and 21, Cycle 1 Day 2, 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 8 | 3 | 1
ratio | 1.51 (47) | 1.36 (79) | 2.11 (6.0) | 1.16 (34) | 1.71 (29) | 1.70 (25) | 2.8 (NA) — Measure dispersion not applicable as only one participant was evaluable.

27. Secondary Outcome: Tmax of Cobimetinib on Cycle 1 Day 1 - Stage 1A All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 15-17
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 9 | 8 | 5
hours | 2.00 [2.0 to 4.0] | 4.00 [2.0 to 6.0] | 2.00 [1.0 to 2.0] | 4.00 [2.0 to 24] | 4.00 [2.0 to 6.0] | 5.00 [2.0 to 24] | 4.00 [2.0 to 6.0]

28. Secondary Outcome: Cmax of Cobimetinib on Cycle 1 Day 1 - Stage 1A All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 15-17
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 9 | 8 | 5
ng/mL | 301 (87) | 137 (66) | 436 (67) | 184 (47) | 275 (72) | 333 (45) | 311 (48)

29. Secondary Outcome: AUC0-24 of Cobimetinib on Cycle 1 Day 1 - Stage 1A All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Days 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 9 | 8 | 5
ng*h/mL | 4950 (80) | 2320 (61) | 5520 (59) | 2620 (50) | 4250 (75) | 5100 (47) | 5090 (45)

30. Secondary Outcome: Tmax of Cobimetinib on Cycle 1 Day 18 - Stage 1A All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 4
hours | 2.00 [2.0 to 4.0] | 2.00 [2.0 to 2.0] | 2.00 [2.0 to 6.0] | 4.00 [2.0 to 6.0] | 4.00 [2.0 to 6.0] | 5.00 [2.0 to 24] | 3.00 [2.0 to 4.0]

31. Secondary Outcome: Cmax of Cobimetinib on Cycle 1 Day 18 - Stage 1A All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 4
ng/mL | 802 (24) | 372 (45) | 616 (39) | 204 (57) | 409 (43) | 475 (86) | 682 (23)

32. Secondary Outcome: AUC0-24 of Cobimetinib on Cycle 1 Day 18 - Stage 1A All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 18, Cycle 1 Day 19
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 4
ng*h/mL | 13400 (18) | 5680 (55) | 9990 (28) | 3060 (50) | 6980 (55) | 7740 (69) | 11100 (23)

33. Secondary Outcome: t1/2 of Cobimetinib on Cycle 1 Day 18 - Stage 1A All Cohorts
Description: Half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 2 | 3 | 3 | 6 | 6 | 2 | 4
hours | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data. | 46.1 [32 to 67] | 47.4 [34 to 63] | 48.8 [37 to 63] | 48 [36 to 72] | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data. | 46.2 [33 to 55]

34. Secondary Outcome: CL/F of Cobimetinib on Cycle 1 Day 18 - Stage 1A All Cohorts
Description: as for outcome 16
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 4
L/hr | 7.49 (18) | 17.6 (55) | 12.5 (28) | 40.9 (50) | 17.9 (55) | 19.4 (69) | 13.6 (23)

35. Secondary Outcome: Accumulation Ratio of Cobimetinib on Cycle 1 Day 18 - Stage 1A All Cohorts
Description: Accumulation ratio was calculated as: AUC0-24 at Cycle 1 Day 18 divided by AUC0-24 at Cycle 1 Day 1.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Days 1 and 18, Cycle 1 Days 2, 19
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 4
ratio | 2.70 (57) | 2.44 (60) | 1.46 (30) | 1.11 (67) | 1.52 (120) | 1.75 (40) | 1.84 (8.1)

36. Secondary Outcome: Tmax of Pictilisib on Cycle 1 Day 1 - Stage 1A All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 15-17
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 9 | 8 | 5
hours | 2.00 [2.0 to 4.0] | 2.00 [2.0 to 2.0] | 2.00 [2.0 to 2.0] | 2.00 [2.0 to 24] | 2.00 [2.0 to 4.0] | 2.00 [0.5 to 6.0] | 4.00 [0.5 to 6.0]

37. Secondary Outcome: Cmax of Pictilisib on Cycle 1 Day 1 - Stage 1A All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 15-17
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 9 | 8 | 5
ng/mL | 547 (80) | 408 (190) | 390 (76) | 367 (61) | 832 (35) | 619 (110) | 514 (81)

38. Secondary Outcome: AUC0-24 of Pictilisib on Cycle 1 Day 1 - Stage 1A All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Days 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 9 | 8 | 5
ng*h/mL | 6900 (62) | 4900 (170) | 3670 (72) | 4280 (48) | 8440 (32) | 5650 (88) | 6680 (53)

39. Secondary Outcome: Tmax of Pictilisib on Cycle 1 Day 18 - Stage 1A All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 4
hours | 2.00 [2.0 to 4.0] | 2.00 [2.0 to 2.0] | 2.00 [0.5 to 2.0] | 2.00 [2.0 to 2.0] | 3.00 [2.0 to 6.0] | 2.00 [0.5 to 6.0] | 3.00 [2.0 to 24]

40. Secondary Outcome: Cmax of Pictilisib on Cycle 1 Day 18 - Stage 1A All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 4
ng/mL | 809 (41) | 709 (71) | 597 (38) | 579 (100) | 833 (49) | 743 (53) | 646 (24)

41. Secondary Outcome: AUC0-24 of Pictilisib on Cycle 1 Day 18 - Stage 1A All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 18, Cycle 1 Day 19
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 4
ng*h/mL | 11300 (21) | 7680 (88) | 6990 (38) | 6120 (110) | 12100 (58) | 8140 (58) | 10100 (44)

42. Secondary Outcome: t1/2 of Pictilisib on Cycle 1 Day 18 - Stage 1A All Cohorts
Description: as for outcome 24
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 2 | 2 | 3 | 1 | 6 | 2 | 2
hours | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data. | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data. | 34.9 [29 to 44] | 36.5 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable. | 38.4 [27 to 52] | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data. | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data.

43. Secondary Outcome: CL/F of Pictilisib on Cycle 1 Day 18 - Stage 1A All Cohorts
Description: as for outcome 16
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 4
L/hr | 11.5 (21) | 23.5 (88) | 18.6 (38) | 29.4 (110) | 20.3 (58) | 22.1 (58) | 24.2 (44)

44. Secondary Outcome: Accumulation Ratio of Pictilisib on Cycle 1 Day 18 - Stage 1A All Cohorts
Description: Accumulation ratio was calculated as: AUC0-24 at Cycle 1 Day 18 divided by AUC0-24 at Cycle 1 Day 1.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Days 1 and 18, Cycle 1 Days 2, 19
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 4
ratio | 1.64 (40) | 1.57 (45) | 1.89 (110) | 1.15 (55) | 1.56 (42) | 1.60 (100) | 1.46 (100)

45. Secondary Outcome: Tmax of Cobimetinib on Cycle 1 Day 1 - Stage 1B All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Day 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3 | 5
hours | 3.00 [2.0 to 6.0] | 2.00 [2.0 to 4.0] | 4.00 [2.0 to 24] | 4.00 [0 to 6.0]

46. Secondary Outcome: Cmax of Cobimetinib on Cycle 1 Day 1 - Stage 1B All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Day 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3 | 5
ng/mL | 55 (160) | 123 (56) | 45.6 (110) | 77.8 (110)

47. Secondary Outcome: AUC0-24 of Cobimetinib on Cycle 1 Day 1 - Stage 1B All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Day 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3 | 1
ng*h/mL | 855 (150) | 1750 (77) | 699 (72) | 2460 (NA) — Measure dispersion not applicable as only one participant was evaluable.

48. Secondary Outcome: Tmax of Cobimetinib on Cycle 1 Day 21 - Stage 1B All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3 | 4
hours | 5.00 [2.0 to 6.0] | 4.00 [2.0 to 6.0] | 2.00 [0 to 6.0] | 6.00 [2.0 to 6.0]

49. Secondary Outcome: Cmax of Cobimetinib on Cycle 1 Day 21 - Stage 1B All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3 | 4
ng/mL | 174 (50) | 232 (120) | 158 (73) | 245 (45)

50. Secondary Outcome: AUC0-24 of Cobimetinib on Cycle 1 Day 21 - Stage 1B All Cohorts
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 2 | 4
ng*h/mL | 3270 (64) | 4320 (150) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data. | 4190 (52)

51. Secondary Outcome: CL/F of Cobimetinib on Cycle 1 Day 21 - Stage 1B All Cohorts
Description: as for outcome 16
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 2 | 4
L/hr | 12.2 (64) | 9.26 (150) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data. | 14.3 (52)

52. Secondary Outcome: Accumulation Ratio of Cobimetinib on Cycle 1 Day 21 - Stage 1B All Cohorts
Description: Accumulation ratio was calculated as: AUC0-24 at Cycle 1 Day 21 divided by AUC0-24 at Cycle 1 Day 1.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Days 1 and 21, Cycle 1 Days 2 and 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 2 | 1
ratio | 3.82 (60) | 2.46 (46) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data. | 1.15 (57)

53. Secondary Outcome: Tmax of Pictilisib on Cycle 1 Day 1 - Stage 1B All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Day 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3 | 5
hours | 2.00 [2.0 to 2.0] | 2.00 [2.0 to 6.0] | 2.00 [2.0 to 24] | 4.00 [2.0 to 6.0]

54. Secondary Outcome: Cmax of Pictilisib on Cycle 1 Day 1 - Stage 1B All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Day 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3 | 5
ng/mL | 527 (67) | 609 (27) | 168 (130) | 363 (64)

55. Secondary Outcome: AUC0-24 of Pictilisib on Cycle 1 Day 1 - Stage 1B All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Day 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3 | 5
ng*h/mL | 5380 (50) | 6540 (20) | 2260 (70) | 4160 (77)

56. Secondary Outcome: Tmax of Pictilisib on Cycle 1 Day 21 - Stage 1B All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3 | 4
hours | 4.00 [0.5 to 6.0] | 2.00 [2.0 to 4.0] | 4.00 [2.0 to 6.0] | 5.00 [0 to 6.0]

57. Secondary Outcome: Cmax of Pictilisib on Cycle 1 Day 21 - Stage 1B All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 3 | 4
ng/mL | 508 (10) | 1010 (27) | 227 (19) | 408 (62)

58. Secondary Outcome: AUC0-24 of Pictilisib on Cycle 1 Day 21 - Stage 1B All Cohorts
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 2 | 4
ng*h/mL | 7000 (12) | 13500 (39) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data. | 5410 (57)

59. Secondary Outcome: CL/F of Pictilisib on Cycle 1 Day 21 - Stage 1B All Cohorts
Description: as for outcome 16
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 2 | 4
L/hr | 18.6 (12) | 13.3 (39) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data. | 33.3 (57)

60. Secondary Outcome: Accumulation Ratio of Pictilisib on Cycle 1 Day 21 - Stage 1B All Cohorts
Description: Accumulation ratio was calculated as: AUC0-24 at Cycle 1 Day 21 divided by AUC0-24 at Cycle 1 Day 1.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Days 1 and 21, Cycle 1 Days 2 and 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 4 | 3 | 2 | 4
ratio | 1.30 (40) | 2.06 (19) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data. | 1.36 (57)

61. Secondary Outcome: Tmax of Cobimetinib on Cycle 1 Day 1 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Groups:
- S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib: Participants with EGFR T790M mutant and EGFR inhibitor-progressing NSCLC received cobimetinib 40 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib: Participants with KRAS NSCLC received cobimetinib 40 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib: Participants with KRAS CRC received cobimetinib 40 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib: Participants with pancreatic adenocarcinoma received cobimetinib 40 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 7 | 9 | 12 | 6
hours | 2.00 [2.0 to 6.0] | 4.00 [2.0 to 24] | 3.00 [2.0 to 6.0] | 4.00 [2.0 to 24]

62. Secondary Outcome: Cmax of Cobimetinib on Cycle 1 Day 1 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 7 | 9 | 12 | 6
ng/mL | 73.8 (38) | 90.7 (87) | 116 (63) | 48.2 (97)

63. Secondary Outcome: AUC0-24 of Cobimetinib on Cycle 1 Day 1 - Stage 2 All Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Days 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 7 | 9 | 12 | 6
ng*h/mL | 1080 (26) | 1330 (100) | 1790 (73) | 700 (84)

64. Secondary Outcome: Tmax of Cobimetinib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 21, Cycle 1 Day 22, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 5 | 8 | 9 | 2
hours | 4.00 [2.0 to 6.0] | 4.00 [2.0 to 6.0] | 2.00 [2.0 to 6.0] | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data.

65. Secondary Outcome: Cmax of Cobimetinib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 21, Cycle 1 Day 22, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 5 | 8 | 9 | 2
ng/mL | 119 (62) | 237 (63) | 254 (120) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

66. Secondary Outcome: AUC0-24 of Cobimetinib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 5 | 8 | 9 | 2
ng*h/mL | 2200 (57) | 4570 (68) | 4700 (120) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

67. Secondary Outcome: t1/2 of Cobimetinib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately. Half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 5 | 8 | 9 | 2
hours | 42.5 [40 to 45] | 51.5 [42 to 83] | 36.0 [28 to 44] | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data.

68. Secondary Outcome: CL/F of Cobimetinib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately. Half-life is the time measured for the plasma concentration to decrease by one half. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 21, Cycle 1 Day 22, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 5 | 8 | 9 | 2
L/hr | 18.2 (57) | 8.76 (68) | 8.52 (120) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

69. Secondary Outcome: Accumulation Ratio of Cobimetinib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately. Accumulation ratio was calculated as: AUC0-24 at Cycle 1 Day 21 divided by AUC0-24 at Cycle 1 Day 1.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Days 1 and 21, Cycle 1 Days 2 and 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 5 | 8 | 9 | 2
ratio | 1.92 (51) | 3.28 (52) | 2.60 (63) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

70. Secondary Outcome: Tmax of Pictilisib on Cycle 1 Day 1 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 7 | 9 | 12 | 6
hours | 2.00 [2.0 to 6.0] | 2.00 [0.5 to 6.0] | 2.00 [0.5 to 4.0] | 4.00 [2.0 to 24]

71. Secondary Outcome: Cmax of Pictilisib on Cycle 1 Day 1 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 7 | 9 | 12 | 6
ng/mL | 298 (52) | 355 (55) | 315 (58) | 253 (90)

72. Secondary Outcome: AUC0-24 of Pictilisib on Cycle 1 Day 1 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Days 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 7 | 9 | 12 | 6
ng*h/mL | 3010 (37) | 3800 (63) | 3210 (59) | 3340 (78)

73. Secondary Outcome: Tmax of Pictilisib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 21, Cycle 1 Day 22, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 4 | 8 | 10 | 2
hours | 4.00 [2.0 to 6.0] | 2.00 [0.5 to 6.0] | 2.00 [2.0 to 4.0] | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data.

74. Secondary Outcome: Cmax of Pictilisib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 21, Cycle 1 Day 22, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 4 | 8 | 10 | 2
ng/mL | 231 (63) | 362 (60) | 369 (66) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

75. Secondary Outcome: AUC0-24 of Pictilisib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: Stage 2 PK data were reported for each indication specific cohort separately.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 21, Cycle 1 Day 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 4 | 8 | 10 | 2
ng*h/mL | 3390 (39) | 5250 (66) | 4580 (56) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

76. Secondary Outcome: t1/2 of Pictilisib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: as for outcome 67
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 21, Cycle 1 Day 22, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 1 | 8 | 10 | 1
hours | 183 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable. | 28.5 [22 to 33] | 26.6 [20 to 37] | 30.9 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable.

77. Secondary Outcome: CL/F of Pictilisib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: as for outcome 68
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 21, Cycle 1 Day 22, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 4 | 8 | 10 | 2
L/hr | 29.5 (39) | 19.1 (66) | 21.8 (56) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

78. Secondary Outcome: Accumulation Ratio of Pictilisib on Cycle 1 Day 21 - Stage 2 Individual Indication Specific Cohorts
Description: as for outcome 69
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Days 1 and 21, Cycle 1 Days 2 and 22
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | S2 EGFR T790M NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS NSCLC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 KRAS CRC: 40 mg Cobimetinib + 100 mg Pictilisib | S2 Pancreatic: 40 mg Cobimetinib + 100 mg Pictilisib
Number analyzed (Participants) | 4 | 8 | 10 | 2
ratio | 0.90 (40) | 1.39 (58) | 1.43 (57) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

79. Secondary Outcome: Tmax of Cobimetinib on Cycle 1 Day 1 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 15-17
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Groups:
- S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib: Participants with EGFR T790M mutant and EGFR inhibitor-progressing NSCLC received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib: Participants with KRAS NSCLC received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib: Participants with KRAS CRC received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib: Participants with pancreatic adenocarcinoma received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib: Participants with KRAS mutant endometrioid carcinoma received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 8 | 12 | 12 | 3
hours | 4.00 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable. | 6.00 [2.0 to 24.0] | 4.00 [2.0 to 24] | 4.00 [2.0 to 24] | 2.00 [2.0 to 4.0]

80. Secondary Outcome: Cmax of Cobimetinib on Cycle 1 Day 1 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 15-17
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 8 | 12 | 12 | 3
ng/mL | 487 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 334 (44) | 256 (130) | 277 (110) | 408 (89)

81. Secondary Outcome: AUC0-24 of Cobimetinib on Cycle 1 Day 1 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 1, Cycle 1 Days 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 8 | 12 | 12 | 3
ng*h/mL | 6560 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 5210 (43) | 4470 (120) | 4090 (120) | 5630 (90)

82. Secondary Outcome: Tmax of Cobimetinib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately. As planned, summary statistics were not derived if fewer than 3 participants had available data; however, if the number of participants analyzed = 1, then the observed data of the single participant was reported as median.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 5 | 8 | 9 | 2
hours | 4.00 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable. | 4.00 [2.0 to 6.0] | 3.00 [2.0 to 6.0] | 4.00 [2.0 to 6.0] | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data.

83. Secondary Outcome: Cmax of Cobimetinib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately. As planned, summary statistics were not derived if fewer than 3 participants had available data; however, if the number of participants analyzed = 1, then the observed data of the single participant was reported as geometric mean.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 5 | 8 | 9 | 2
ng/mL | 587 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 502 (16) | 469 (40) | 393 (44) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

84. Secondary Outcome: AUC0-24 of Cobimetinib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: as for outcome 83
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 5 | 8 | 9 | 2
ng*h/mL | 9560 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 7920 (16) | 7390 (32) | 5790 (46) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

85. Secondary Outcome: t1/2 of Cobimetinib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately. Half-life is the time measured for the plasma concentration to decrease by one half. As planned, summary statistics were not derived if fewer than 3 participants had available data; however, if the number of participants analyzed = 1, then the observed data of the single participant was reported as geometric mean.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 5 | 8 | 9 | 2
hours | 37.7 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable. | 38.6 [33 to 42] | 50.2 [35 to 89] | 42.6 [27 to 64] | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data.

86. Secondary Outcome: CL/F of Cobimetinib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. As planned, summary statistics were not derived if fewer than 3 participants had available data; however, if the number of participants analyzed = 1, then the observed data of the single participant was reported as geometric mean.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 5 | 8 | 9 | 2
L/hr | 13.1 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 15.8 (16) | 16.9 (32) | 21.6 (46) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

87. Secondary Outcome: Accumulation Ratio of Cobimetinib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately. Accumulation ratio was calculated as: AUC0-24 at Cycle 1 Day 21 divided by AUC0-24 at Cycle 1 Day 1. As planned, summary statistics were not derived if fewer than 3 participants had available data; however, if the number of participants analyzed = 1, then the observed data of the single participant was reported as geometric mean.
Time Frame: Pr-C dose, 0.5, 2, 4, 6 hours Po-C dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 5 | 8 | 9 | 2
ng*h/mL | 1.46 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 1.43 (51) | 1.89 (94) | 1.72 (83) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

88. Secondary Outcome: Tmax of Pictilisib on Cycle 1 Day 1 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 15-17
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 8 | 12 | 12 | 3
hours | 2.00 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable. | 2.00 [0.5 to 6.0] | 2.00 [0.5 to 6.0] | 2.00 [0.5 to 24] | 4.00 [2.0 to 6.0]

89. Secondary Outcome: Cmax of Pictilisib on Cycle 1 Day 1 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Days 2, 8, 15-17
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 8 | 12 | 12 | 3
ng/mL | 714 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 265 (140) | 289 (100) | 393 (90) | 369 (35)

90. Secondary Outcome: AUC0-24 of Pictilisib on Cycle 1 Day 1 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 1, Cycle 1 Days 2
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 8 | 12 | 12 | 3
ng*h/mL | 8050 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 3380 (100) | 3310 (76) | 4030 (88) | 4500 (16)

91. Secondary Outcome: Tmax of Pictilisib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: as for outcome 83
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 5 | 8 | 9 | 2
hours | 2.00 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable. | 2.00 [2.0 to 24] | 2.00 [0.5 to 4.0] | 2.00 [2.0 to 6.0] | NA [NA to NA] — As planned, summary statistics were not derived if fewer than 3 participants had available data.

92. Secondary Outcome: Cmax of Pictilisib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: as for outcome 83
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 5 | 8 | 9 | 2
ng/mL | 412 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 518 (67) | 520 (84) | 334 (83) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

93. Secondary Outcome: AUC0-24 of Pictilisib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: as for outcome 83
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 5 | 8 | 9 | 2
ng*h/mL | 6300 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 6310 (31) | 5930 (73) | 3990 (74) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

94. Secondary Outcome: t1/2 of Pictilisib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: Stage 2A PK data were reported for each indication specific cohort separately. Half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 0 | 5 | 8 | 9 | 1
hours |  | 44.6 [28 to 66] | 58.2 [40 to 83] | 37.8 [29 to 50] | 30.3 [NA to NA] — Measure dispersion not applicable as only one participant was evaluable.

95. Secondary Outcome: CL/F of Pictilisib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: as for outcome 86
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 5 | 8 | 9 | 2
L/hr | 28.6 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 28.5 (31) | 30.3 (73) | 45.1 (74) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

96. Secondary Outcome: Accumulation Ratio of Pictilisib on Cycle 1 Day 18 - Stage 2A Individual Indication Specific Cohorts
Description: as for outcome 87
Time Frame: Pr-P dose, 0.5, 2, 4, 6 hours Po-P dose on Cycle 1 Day 18, Cycle 1 Day 19, Cycle 2 Days 1, 15, 21
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | S2A EGFR T790M NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS NSCLC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A KRAS CRC: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Pancreatic: 125 mg Cobimetinib + 180 mg Pictilisib | S2A Endometrioid: 125 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 1 | 5 | 8 | 9 | 2
ng*h/mL | 0.78 (NA) — Measure dispersion not applicable as only one participant was evaluable. | 1.61 (110) | 1.90 (50) | 1.03 (84) | NA (NA) — As planned, summary statistics were not derived if fewer than 3 participants had available data.

97. Secondary Outcome: Number of Participants With Best Overall Response - Dose Escalation Stages 1, 1A and 1B
Description: Tumor response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) = disappearance of all target and non-target lesions. Partial Response (PR) = at least 30 percent (%) decrease in sum of the longest diameter of measured lesions taking as reference the baseline sum of the longest diameter. Progressive disease (PD) = at least 20% increase in the sum of the longest diameter of measured lesions taking as reference the smallest sum of the longest diameter since treatment start or appearance of one or more new lesions. Stable disease (SD) = neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter since treatment start.
Time Frame: Up to 30 days after last dose (last dose = up to Cycle 15, cycle length = 28 days)
Population: Safety-evaluable population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: participants
Groups:
- S1 C4/S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib: Participants received cobimetinib 40 mg capsules and pictilisib 100 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. This arm included participants from S1 C4 as well as S2 expansion cohort.
- S1A CD/S2A Expension: 125 mg Cobimetinib + 180 mg Pictilisib: Participants received cobimetinib 125 mg capsules on Days 1, 4, 8, 11, 15, and 18 and pictilisib 180 mg capsules from Days 1 to 21 and then 7 days off study drugs from Days 22 to 28 in continuous 28-day cycles. Treatment continued until disease progression, unacceptable toxicity, or any other discontinuation criterion was met. This arm included participants form S1A CD as well as S2A expansion cohort.
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4/S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD/S2A Expension: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 2 | 3 | 3 | 31 | 10 | 8 | 1 | 2 | 3 | 4 | 35 | 7 | 6 | 3 | 4 | 3 | 3 | 3
participants
  PR | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SD | 2 | 2 | 1 | 15 | 5 | 3 | 1 | 0 | 2 | 3 | 16 | 5 | 2 | 0 | 1 | 1 | 0 | 1
  PD | 0 | 1 | 2 | 16 | 5 | 4 | 0 | 2 | 1 | 0 | 17 | 1 | 4 | 3 | 3 | 2 | 3 | 2
  Unable to Evaluate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

98. Secondary Outcome: Duration of Objective Response - Dose Escalation Stages 1, 1A and 1B
Description: Duration of objective response was defined as the time from first occurrence of a documented objective response (CR or PR) until the time of disease progression, as determined by investigator review of tumor assessments using RECIST, or death from any cause during the study (within 30 days after the last dose of study treatment). CR = disappearance of all target and non-target lesions. PR = at least 30 % decrease in sum of the longest diameter of measured lesions taking as reference the baseline sum of the longest diameter. PD = at least 20% increase in the sum of the longest diameter of measured lesions taking as reference the smallest sum of the longest diameter since treatment start or appearance of one or more new lesions.
Time Frame: Up to 30 days after last dose (last dose = up to Cycle 15, cycle length = 28 days)
Population: Data for this outcome measure was not collected as per changes in planned analysis.
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4/S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD/S2A Expension: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

99. Secondary Outcome: Progression-Free Survival (PFS) - Dose Escalation Stages 1, 1A and 1B
Description: PFS was the time from study treatment initiation to the first occurrence of disease progression, as determined by investigator review of tumor assessments using RECIST, or death from any cause during the study (within 30 days after the last dose of study treatment). PD = at least 20% increase in the sum of the longest diameter of measured lesions taking as reference the smallest sum of the longest diameter since treatment start or appearance of one or more new lesions.
Time Frame: Up to 30 days after last dose (last dose = up to Cycle 15, cycle length = 28 days)
Population: Data for this outcome measure was not collected as per changes in planned analysis.
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4/S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD/S2A Expension: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose (last dose = up to Cycle 15, cycle length = 28 days)
Description: Safety evaluable population.
Arm/Group | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib | S1 C4/S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib | S1A CD/S2A Expension: 125 mg Cobimetinib + 180 mg Pictilisib | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 1/3 | 25/43 | 6/11 | 6/10 | 2/4 | 2/3 | 2/3 | 3/4 | 28/52 | 4/9 | 5/8 | 3/5 | 0/4 | 0/3 | 0/3 | 2/5
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 42/43 | 11/11 | 10/10 | 4/4 | 3/3 | 3/3 | 4/4 | 52/52 | 9/9 | 8/8 | 5/5 | 4/4 | 3/3 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib (N=4) | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib (N=3) | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib (N=3) | S1 C4/S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib (N=43) | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib (N=11) | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib (N=10) | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib (N=4) | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib (N=3) | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib (N=3) | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib (N=4) | S1A CD/S2A Expension: 125 mg Cobimetinib + 180 mg Pictilisib (N=52) | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib (N=9) | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib (N=8) | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib (N=5) | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib (N=4) | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib (N=3) | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib (N=3) | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colititis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ercherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitits (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | S1 C1: 20 mg Cobimetinib + 80 mg Pictilisib (N=4) | S1 C2: 20 mg Cobimetinib + 100 mg Pictilisib (N=3) | S1 C3: 40 mg Cobimetinib + 80 mg Pictilisib (N=3) | S1 C4/S2 Expansion: 40 mg Cobimetinib + 100 mg Pictilisib (N=43) | S1 C5: 40 mg Cobimetinib + 130 mg Pictilisib (N=11) | S1 C6: 60 mg Cobimetinib + 100 mg Pictilisib (N=10) | S1 C6A: 80 mg Cobimetinib + 100 mg Pictilisib (N=4) | S1A CA: 100 mg Cobimetinib + 130 mg Pictilisib (N=3) | S1A CB: 100 mg Cobimetinib + 180 mg Pictilisib (N=3) | S1A CC: 125 mg Cobimetinib + 130 mg Pictilisib (N=4) | S1A CD/S2A Expension: 125 mg Cobimetinib + 180 mg Pictilisib (N=52) | S1A CE: 125 mg Cobimetinib + 245 mg Pictilisib (N=9) | S1A CF: 150 mg Cobimetinib + 180 mg Pictilisib (N=8) | S1A CG: 150 mg Cobimetinib + 245 mg Pictilisib (N=5) | S1B CAX: 40 mg Cobimetinib + 130 mg Pictilisib (N=4) | S1B CBX: 40 mg Cobimetinib + 180 mg Pictilisib (N=3) | S1B CCX: 60 mg Cobimetinib + 130 mg Pictilisib (N=3) | S1B CDX: 60 mg Cobimetinib + 180 mg Pictilisib (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 5 | 0 | 3 | 0 | 2 | 1 | 0 | 7 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 0 | 2 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Photophobia (Eye disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Visual impairment (Eye disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 16 | 2 | 1 | 0 | 1 | 0 | 1 | 16 | 3 | 2 | 0 | 0 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 3 | 39 | 9 | 8 | 4 | 2 | 3 | 4 | 44 | 8 | 7 | 4 | 3 | 2 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 6 | 2 | 2 | 0 | 0 | 2 | 1 | 5 | 0 | 2 | 1 | 0 | 1 | 0 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 8 | 0 | 2 | 0 | 0 | 0 | 2 | 13 | 0 | 2 | 1 | 0 | 1 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2 | 3 | 25 | 6 | 6 | 3 | 1 | 3 | 3 | 36 | 7 | 7 | 3 | 1 | 2 | 1 | 5
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 11 | 1 | 3 | 2 | 1 | 3 | 2 | 12 | 4 | 1 | 1 | 0 | 0 | 1 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 2 | 27 | 5 | 8 | 3 | 2 | 0 | 4 | 32 | 5 | 6 | 3 | 0 | 3 | 1 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 2 | 3 | 1 | 1 | 1 | 0 | 0 | 1 | 6 | 3 | 1 | 1 | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 1 | 1 | 26 | 5 | 5 | 3 | 1 | 2 | 2 | 29 | 6 | 7 | 3 | 3 | 1 | 2 | 2
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localized oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 7 | 4 | 2 | 0 | 1 | 1 | 2 | 8 | 2 | 0 | 2 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 11 | 4 | 3 | 1 | 1 | 1 | 2 | 16 | 3 | 1 | 1 | 0 | 1 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitits (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Penile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 5 | 1 | 1 | 1 | 0 | 1 | 1 | 3 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site rash (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 4 | 2 | 4 | 1 | 0 | 1 | 2 | 3 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 0 | 5 | 3 | 3 | 0 | 0 | 1 | 2 | 6 | 2 | 2 | 2 | 2 | 0 | 0 | 0
Blood creatine phosphokinase mb increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haermatocrit decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 9 | 1 | 2 | 0 | 0 | 1 | 2 | 6 | 2 | 3 | 2 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 16 | 3 | 5 | 1 | 1 | 3 | 4 | 21 | 3 | 5 | 2 | 2 | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 8 | 2 | 5 | 2 | 1 | 1 | 0 | 9 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 9 | 2 | 2 | 1 | 0 | 0 | 0 | 10 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 1 | 4 | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 8 | 0 | 1 | 0 | 0 | 1 | 0 | 6 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consiousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 10 | 1 | 1 | 1 | 0 | 1 | 1 | 9 | 2 | 3 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 16 | 3 | 2 | 0 | 2 | 3 | 1 | 16 | 3 | 5 | 2 | 2 | 2 | 1 | 1
Headache (Nervous system disorders) | 2 | 1 | 0 | 7 | 2 | 1 | 0 | 0 | 0 | 0 | 7 | 2 | 0 | 4 | 0 | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trigeminal palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 9 | 3 | 2 | 0 | 0 | 1 | 3 | 8 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 8 | 3 | 2 | 0 | 0 | 1 | 0 | 13 | 3 | 0 | 0 | 0 | 0 | 0 | 2
Dysnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 8 | 1 | 4 | 0 | 0 | 0 | 1 | 15 | 2 | 4 | 1 | 2 | 1 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6 | 0 | 3 | 0 | 2 | 0 | 1 | 5 | 3 | 1 | 2 | 0 | 1 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 6 | 2 | 0 | 0 | 1 | 1 | 2 | 7 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 9 | 8 | 2 | 3 | 0 | 3 | 2 | 19 | 3 | 1 | 0 | 1 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 16 | 3 | 3 | 0 | 1 | 0 | 1 | 12 | 4 | 3 | 4 | 0 | 1 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin maceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Wound drainage (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated prior to the initiation of Stage 2B and as per changes in planned analysis the data for duration of objective response and PFS were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.